CLINICAL TRIAL: NCT06127719
Title: The Effects of Surgical Wait Time on Function, Pain and Health Related Quality of Life in Patients Awaiting Knee Arthroplasty: a Prospective Multicenter Cohort Study
Brief Title: The Effects of Surgical Wait Time for Knee Arthroplasty Quality of Life in Patients Awaiting Knee Arthroplasty
Acronym: SIT'NWAIT
Status: Recruiting | Type: Observational
Sponsor: Dijklander Ziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: DOC 23-023
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee arthroplasty; surgical waiting time; waiting list; knee pain; total knee arthroplasy; partial knee arthroplasty; knee function; quality of life; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient on the waiting list for knee arthroplasty: adult patient on the waiting list for knee arthroplasty
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — before surgery, patients are asked to fill out the questionnaires as stated in the outcome measures paragraph

SUMMARY:
This study prospectively evaluates the effect of surgical wait time on knee function, pain and quality of life in patients waiting for knee arthroplasty (TKA or PKA)

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common condition, leading to pain and disability. The knee is the most affected joint, accounting for almost 80 percent of the total prevalence of OA. The pooled global prevalence of knee OA is 22.9% in individuals aged 40 and over. Correspondingly, there are around 654.1 million individuals with knee OA in 2020 worldwide. The number of people affected with symptomatic knee OA is likely to increase because of the aging population and the obesity epidemic.

Pain is the most important symptom in knee OA. It is intermittent, typically weight bearing and progressive over time. Additional symptoms are crepitus, swelling and morning stiffness. The knee is often swollen and has diminished range of motion (ROM). Not only does OA lead to functional disability, but also influences social participation and quality of life.

Knee OA is a progressive disease, which requires continuous management. Treatment consists of conservative as well as invasive treatments, as described in national and international guidelines. First line treatments are patient education, physical therapy, weight loss, different pharmacological treatments and intra-articular steroid injections. More advanced OA may require surgery. Knee arthroplasty, (total knee arthroplasty (TKA) or partial knee arthroplasty (PKA)) can provide excellent pain relief, remarkable deformity correction, and satisfactory functional recovery.

Since the beginning of the covid19 pandemic, surgeons have been asked to only perform essential surgeries in order to preserve healthcare resources. This has led to an increase in patients on the waiting list, resulting in unusually high wait times. Despite the decrease in covid related healthcare consumption, waiting times are yet to return to pre-covid duration. Currently, time to surgery in our hospital is approximately 7 months as opposed to 2-3 months pre-covid.

Long wait times may be a substantial burden for patients. There have been reports of worsening pain, deterioration in quality of life and increased opioid use and frailty. The effects on pain catastrophizing, fear and anxiety have not yet been studied.

It is important to better understand the effects of long surgical wait times on pre-operative knee function, pain and quality of life as well as to investigate how this effects outcome after surgery.

ELIGIBILITY:
Inclusion Criteria:

* on the waiting list for partial or total knee arthroplasty
* written informed consent

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients on the waiting list for knee arthroplasty (TKA or PKA).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Knee function measured with the Oxford knee score (OKS) | Baseline, before surgery
  This questionnaire consists of 12 items, which are divided into disease-specific and generic questions. Scores can range from 0 - 48, lower scores indicate more functional limitations and pain.

SECONDARY OUTCOMES:
numeric rating scale for pain (NRS) | baseline, before surgery, 6 and 12 months postoperatively
  This scale consists of 11 numbers from 0-10, where 0 means no pain at all and 10 is the most pain imaginable. The patient should circle the number that best represents the severity of pain experienced over the past week
Health related quality of life with the euroqol 5 dimensions (EQ-5D-5L) | baseline, before surgery, 6 and 12 months postoperatively
  The EQ-5D is a questionnaire that scores five health dimensions (mobility, self-care, daily activities, pain/discomfort and anxiety/depression). Patient must indicate their health status: no problems, slight problems, moderate problems, severe problems, extreme problems.
Hospital anxiety and depression scale (HADS) | baseline, before surgery, 6 and 12 months postoperatively
  This is a short questionnaire that is easy to use. The scale examines feelings in the past week and consists of an anxiety scale and a depression scale with both 7 items. The higher a patient scores on this questionnaire, the more complaints one experiences.
Pain catastrophizing scale (PCS) | baseline, before surgery, 6 and 12 months postoperatively
  This self-assessment questionnaire consists of 13 statements that contain a number of thoughts and feelings that one may experience having pain. The items are divided into the categories rumination, magnification and helplessness, with each item scored on a 5-point scale. The sum of scores ranges from 0 - 52, with higher scores indicating higher levels of catastrophizing.

OTHER OUTCOMES:
medical consumption questionnaire (iMCQ) | before surgery
  The iMCQ includes questions related to frequently occurring contacts with health care providers. Reference is made to healthcare consumption due to illness, disability or psychiatric problems, without specifying a particular disease. Healthcare consumption in the preceding 13 weeks is applicable.
Knee function measured with the Oxford knee score (OKS) | 6 and 12 months postoperatively
  This questionnaire consists of 12 items, which are divided into disease-specific and generic questions. Scores can range from 0 - 48, lower scores indicate more functional limitations and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gezina TM Oei, dr, Study Director — Department of anesthesiology Dijklander Hospital
Locations (1):
- Dijklander Hospital, Hoorn, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Background] Bertrix L, Lakhal M, Timour Chah Q, Lang J, Foussat C, Faucon G. [Caudal anesthesia by lidocaine in children. Diffusion in the blood and possible cardiac effects]. Therapie. 1985 Jul-Aug;40(4):225-9. No abstract available. French. PMID 4024017
- [Background] Bunt CW, Jonas CE, Chang JG. Knee Pain in Adults and Adolescents: The Initial Evaluation. Am Fam Physician. 2018 Nov 1;98(9):576-585. PMID 30325638
- [Background] Hunter DJ, Bierma-Zeinstra S. Osteoarthritis. Lancet. 2019 Apr 27;393(10182):1745-1759. doi: 10.1016/S0140-6736(19)30417-9. PMID 31034380
- [Background] Bruyere O, Honvo G, Veronese N, Arden NK, Branco J, Curtis EM, Al-Daghri NM, Herrero-Beaumont G, Martel-Pelletier J, Pelletier JP, Rannou F, Rizzoli R, Roth R, Uebelhart D, Cooper C, Reginster JY. An updated algorithm recommendation for the management of knee osteoarthritis from the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Semin Arthritis Rheum. 2019 Dec;49(3):337-350. doi: 10.1016/j.semarthrit.2019.04.008. Epub 2019 Apr 30. PMID 31126594
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] van Geene AR, Saris DB, Custers RJ. [Pain following primary total knee replacement: causes, diagnosis and treatment]. Ned Tijdschr Geneeskd. 2015;159:A8445. Dutch. PMID 26395566
- [Background] Bedard NA, Elkins JM, Brown TS. Effect of COVID-19 on Hip and Knee Arthroplasty Surgical Volume in the United States. J Arthroplasty. 2020 Jul;35(7S):S45-S48. doi: 10.1016/j.arth.2020.04.060. Epub 2020 Apr 24. PMID 32381441
- [Background] Clement ND, Scott CEH, Murray JRD, Howie CR, Deehan DJ; IMPACT-Restart Collaboration. The number of patients "worse than death" while waiting for a hip or knee arthroplasty has nearly doubled during the COVID-19 pandemic. Bone Joint J. 2021 Apr;103-B(4):672-680. doi: 10.1302/0301-620X.103B.BJJ-2021-0104.R1. Epub 2021 Mar 23. PMID 33752468
- [Background] Clement ND, Wickramasinghe NR, Bayram JM, Hughes K, Oag E, Heinz N, Fraser E, Jefferies JG, Dall GF, Ballantyne A, Jenkins PJ. Significant deterioration in quality of life and increased frailty in patients waiting more than six months for total hip or knee arthroplasty : a cross-sectional multicentre study. Bone Joint J. 2022 Nov;104-B(11):1215-1224. doi: 10.1302/0301-620X.104B11.BJJ-2022-0470.R2. PMID 36317352
- [Background] Farrow L, Gardner WT, Tang CC, Low R, Forget P, Ashcroft GP. Impact of COVID-19 on opioid use in those awaiting hip and knee arthroplasty: a retrospective cohort study. BMJ Qual Saf. 2023 Aug;32(8):479-484. doi: 10.1136/bmjqs-2021-013450. Epub 2021 Sep 14. PMID 34521769
- [Background] Henry EB, Barry LE, Hobbins AP, McClure NS, O'Neill C. Estimation of an Instrument-Defined Minimally Important Difference in EQ-5D-5L Index Scores Based on Scoring Algorithms Derived Using the EQ-VT Version 2 Valuation Protocols. Value Health. 2020 Jul;23(7):936-944. doi: 10.1016/j.jval.2020.03.003. Epub 2020 May 14. PMID 32762996
- See also: Dutch national guideline for non-traumatic knee complaints — https://richtlijnen.nhg.org/standaarden/niet-traumatische-knieklachten
- See also: Dutch national guideline for knee arthroplasty — https://richtlijnendatabase.nl/richtlijn/totale_knieprothese/startpagina_-_totale_knieprothese_tkp.html